CLINICAL TRIAL: NCT00843986
Title: A Phase-3b, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Safety and Efficacy of Conivaptan in Symptomatic Acute Decompensated Heart Failure (ADHF) Subjects With Hyponatremia
Brief Title: Safety and Efficacy of Conivaptan in Hyponatremic Patients With Symptomatic Acute Decompensated Heart Failure (ADHF)
Acronym: CONVERT-H
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The clinical study has been terminated based on difficulties to enroll eligible subjects per protocol inclusion and exclusion criteria.
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 087-CL-301
Record Dates: First submitted 2009-02-11; First posted 2009-02-13 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Hyponatremia; Acute Decompensated Heart Failure
Keywords: hyponatremia; euvolemic hyponatremia; hypervolemic hyponatremia; acute decompensated heart failure; conivaptan; Vaprisol
MeSH Terms: conditions — Hyponatremia | interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching loading dose and continuous intravenous infusion for 48 hours
  Interventions: Drug: placebo
- Conivaptan (Experimental): 20mg loading dose followed by a 20mg/ day continuous intravenous infusion for 48 hours
  Interventions: Drug: conivaptan

INTERVENTIONS:
Drug: conivaptan — Premix bag
  Other Names: Vaprisol; YM087
  Arms: Conivaptan
Drug: placebo — Premix bag
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and effectiveness of Conivaptan, a vasopressin antagonist, in the treatment of hyponatremic subjects having symptomatic acute decompensated heart failure (ADHF).

DETAILED DESCRIPTION:
Subjects will be recruited from the Emergency Department. It is expected that subjects will be treated according to the institution's accepted conventional therapy protocol for the treatment of ADHF. Therapy may also include the use of loop diuretics for the relief of pulmonary congestion and maintenance of adequate urine output.

ELIGIBILITY:
Inclusion Criteria:

* Presents to emergency department with documented history of CHF and symptomatic ADHF, will be treated for ADHF, and primary reason for admission to the hospital is ADHF
* Dyspnea at rest or with minimal exertion and must have moderate shortness of breath (SOB) in any of the first three Provocative Dyspnea Assessment positions
* Severe pulmonary congestion as evidenced by jugular venous distention or lower extremity/sacral edema or rales upon chest auscultation or chest x-ray.
* BNP > 400 or NT-pro BNP > 1500 drawn during Screening
* Systolic blood pressure >= 100 mmHg to < 180 mmHg at time of start of study drug
* Serum sodium value >= 115 mEq/L (115 mmol/L) and < 135 mEq/L (135 mmol/L) during Screening

Exclusion Criteria:

* Clinical evidence of volume depletion
* Active ongoing acute coronary syndrome or acute ST segment elevation myocardial infarction (or has experienced a myocardial infarction within 30 days of Screening)
* In cardiogenic shock
* Calculated creatinine clearance < 30 mL/min/1.73 m2 as estimated by the Modification of Diet in Renal Disease (MDRD) equation, has received intravenous (IV) contrast agent within 72 hours prior to randomization or is expected to receive IV contrast agent within the first 72 hours of study participation
* Ultrafiltration within the past 72 hours.
* Currently using or expected to use inotropic therapy
* Cardiac bypass grafts in the past 60 days
* Cerebrovascular accident in the past 30 days
* Uncontrolled brady- or ventricular tachyarrhythmias requiring emergent pacemaker placement or treatment
* Hemodynamically significant uncorrected primary cardiac valvular disease or hypertrophic cardiomyopathy
* Untreated severe hypothyroidism, hyperthyroidism or adrenal insufficiency based on medical history
* ALT or AST elevations > 5 times upper limit of normal
* Biliary liver cirrhosis, history or presence of severe hepatic encephalopathy, ascites, esophageal variceal bleeding within the past three months, severe portal hypertension or surgical portosystemic shunt.
* Received any organ transplant, clinical diagnosis of pneumonia, symptomatic hyponatremia requiring urgent intervention or any concurrent illness which, in the opinion of the investigator, may interfere with treatment or evaluation of safety
* Pregnant or lactating
* Currently using vasopressin, oxytocin or desmopressin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (3):
- India (3):
  - Hyderabaad
  - Karnāl
  - New Delhi

REFERENCES:
- See also: Link to Prescribing Information — http://www.astellas.us/docs/vaprisol.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Conivaptan
Started | 3 | 6
Completed Treatment (Infusion) | 2 | 6
Completed | 2 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Conivaptan | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (13.05) | 65.8 (7.78) | 62.8 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 5 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Renal Function From Baseline at 72 Hours Assessed by Calculated Creatinine Clearance (MDRD Equation)
Description: MDRD = Modification of Diet in Renal Disease
  The MDRD equation is a standard calculation for estimated glomerular filtration rate.
  Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Baseline and 72 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Assessment of Dyspnea at 24 Hours as Determined by a 7-point Likert Scale
Description: Dyspnea is defined as the sensation of uncomfortable or difficult breathing.
  Changes in Dyspnea were assessed using the following 7-point scale: 1-Markedly worse; 2-Moderately worse; 3-Mildly worse; 4-No change; 5-Mildly improved; 6-Moderately improved; 7-Markedly better/improved.
  Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: 24 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Renal Function From Baseline at Hours 24, 48 and 72 as Assessed by Urine Creatinine Clearance
Description: Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Baseline, 24 Hours, 48 Hours and 72 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Renal Function From Baseline at Hours 24, 48 and Day 9 (or Day of Discharge) as Assessed by Serum Creatinine Concentration and Calculated Creatinine Clearance
Description: Calculated creatinine clearance is only calculated through hour 72 using the MDRD equation.
  MDRD = Modification of Diet in Renal Disease
  The MDRD equation is a standard calculation for estimated glomerular filtration rate.
  Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Baseline, 24 Hours, 48 Hours and Day 9
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Use of Rescue Therapy or Other Intervention (Including Dialysis) Because of Worsening Renal Function
Description: Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Day 9
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Termination of Study Drug Due to an Adverse Event or Intolerability
Description: Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: 48.5 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Assessment of Dyspnea at Baseline, Hours 6, 12, 24 and 48 Using a Relative Dyspnea Assessment
Description: Dyspnea is defined as the sensation of uncomfortable or difficult breathing.
  Changes in Dyspnea were assessed using the following 7-point Likert scale:
  1-Markedly worse; 2-Moderately worse; 3-Mildly worse; 4-No change; 5-Mildly improved; 6-Moderately improved; 7-Markedly better/improved.
  Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Baseline, 6 Hours, 12 Hours, 24 Hours and 48 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Assessment of Dyspnea at Baseline, Hours 6, 12, 24 and 48 Using a Provocative Dyspnea Assessment
Description: Dyspnea is defined as the sensation of uncomfortable or difficult breathing.
  The Provocative Dyspnea Assessment assesses dyspnea and changes in dyspnea from Baseline on a 5-point Likert scale at 5 different positions and assigns a Dyspnea Severity Score that ranges from 1 (worst severity) to 25 (least severity).
  Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Baseline, 6 Hours, 12 Hours, 24 Hours and 48 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Body Weight at Hours 24, 48 and 72 and Days 6 and 9 (or Day of Discharge)
Description: Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: Baseline, 24 Hours, 48 Hours, 72 Hours, Day 6 and Day 9
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Total Loop Diuretic Use Through 48 Hours
Description: Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: 48 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Total Urine Output at Hours 6, 12, 24, 48 and 72
Description: Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.
Time Frame: 6 Hours, 12 Hours, 24 Hours, 48 Hours and 72 Hours
Population: Study was terminated - assessment of this Outcome Measure was not performed.
Arm/Group | Placebo | Conivaptan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event collection will begin at the start of study drug infusion and continue through Day 9/ Day of Discharge.
Description: Treatment Emergent Adverse Events are reported and are defined as Adverse Events recorded during the treatment and follow-up periods of the study.
Arm/Group | Placebo | Conivaptan
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6
Other Adverse Events (participants affected / at risk) | 1/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Conivaptan (N=6)
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Conivaptan (N=6)
Atrial flutter (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Infusion site erythema (General disorders) | 0 | 3
Infusion site pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated because of difficulties in enrolling eligible patients per the protocol inclusion and exclusion criteria.

Outcome Measures were not analyzed due to the abbreviated enrollment at early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.